CLINICAL TRIAL: NCT06905041
Title: The Impact of Preoperative Anemia on Postoperative Outcomes in Liver Resection: A Propensity Score Matching Analysis
Brief Title: Preoperative Anemia Affected to Postoperative Outcomes in Liver Resection
Status: Not yet recruiting | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Warangkana Lapisatepun, Faculty of Medicine, Chiang Mai University, Chiang Mai University
Other Study IDs: ANE-2568-0141
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Liver Resection; Anemia; Postoperative Mortality and Morbidity
Keywords: Preoperative anemia, liver resection, posteoperative complication
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anemia group: The patients who had preoperative anemia (hemoglobin levels < 12 g/dL in female and < 13 g/dL in male) before liver resection
- No anemia group: The patients who did not have preoperative anemia before liver resection.

SUMMARY:
To assess the impact of preoperative anemia on postoperative outcomes in patients undergoing liver resection

DETAILED DESCRIPTION:
Globally, anemia affects approximately 33% of the population, with nearly 50% of cases attributed to iron deficiency. In Thailand, anemia remains a significant public health issue, with prevalence rates of 24% among women of reproductive age, 23.8% among nonpregnant women, and 32.2% among pregnant women. Iron deficiency anemia (IDA) is the leading and most common cause of anemia worldwide, and it is highly prevalent in Thailand. Moreover, the situation in Thailand is often exacerbated by the widespread incidence of thalassemia and hemoglobinopathies, with 30% to 40% of the population carrying thalassemia genes.

According to the World Health Organization (WHO), anemia is defined as a hemoglobin concentration of less than 12 g/dL in nonpregnant women and less than 13 g/dL in men. The prevalence of preoperative anemia among surgical patients has been reported to be between 32% and 48%. Preoperative anemia is one of the most common medical conditions encountered in surgical patients, with a prevalence ranging from 20% to 45% depending on the type of surgery. Specifically, in hepato-pancreato-biliary (HPB) surgery, 16.9% to 32.8% of patients present with anemia prior to surgery.

Preoperative anemia is a well-established predictor of the need for perioperative blood transfusions in liver resection, as supported by multiple studies. Perioperative allogeneic blood transfusions are associated with numerous adverse outcomes, both short-term and long-term. These include transfusion reactions, increased rates of postoperative infections, cardiopulmonary and thromboembolic events, prolonged mechanical ventilation, re-operations, extended hospital and ICU stays, elevated postoperative morbidity, increased tumor recurrence, reduced disease-specific survival, and decreased overall survival.

A large retrospective study reported a prevalence of preoperative anemia at 32.8%, which was associated with higher rates of postoperative major morbidities and mortality. After adjusting for confounding factors-such as age, type of liver resection, ASA classification, preoperative laboratory results, comorbidities, functional status, and diagnosis-patients with preoperative anemia were found to have a 21% higher risk of developing major morbidities within 30 days (adjusted odds ratio 1.21, 1.09-1.33). These morbidities included organ space infections, sepsis, septic shock, prolonged postoperative ventilator use (>48 hours), unplanned reintubation, pneumonia, and acute kidney injury requiring dialysis. However, preoperative anemia was not associated with increased postoperative mortality in liver resection (adjusted odds ratio 0.88, 0.66-1.16).

Furthermore, a retrospective study involving 4,170 patients demonstrated that preoperative anemia was associated with an increased risk of major postoperative complications compared to patients without anemia (24% versus 19%). After adjusting for confounders, including age, sex, race, obesity, extent of liver resection, comorbidities, functional status, and clinical and biochemical markers of liver dysfunction and portal hypertension, preoperative anemia was linked to a threefold increased risk of blood transfusion, a twofold increased risk of prolonged hospitalization, and higher healthcare costs in anemic patients. These findings suggest that anemia significantly impacts resource utilization in liver resection.

In a broader context, a study involving 227,425 patients from the ACS-NSQIP database who underwent major non-cardiac surgery reported that 30.4% of patients had preoperative anemia. The results showed that preoperative anemia was associated with increased morbidity and mortality within 30 days, even after adjusting for several known risk factors, including transfusions. Despite this evidence, there are limited studies specifically evaluating the impact of preoperative anemia on outcomes in specific surgeries, particularly liver resection.

The findings of this study could enhance physicians' understanding of the impact of preoperative anemia on postoperative outcomes, emphasizing the importance of its evaluation and treatment. Therefore, the assessment and management of preoperative anemia are essential components of patient blood management in liver resection. Proper assessment and timely intervention could mitigate associated risks and improve surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All genders, age 20 to 75 years old who undergoing elective liver resection
* American Society of Anesthesiologists (ASA) physical status classification of I-III

Exclusion Criteria:

* Living donor liver resection

Withdrawal criteria:

* Unresectable tumor
* Cardiac arrest during operation

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent elective liver resection in setting hospital during January, 2006 to December, 2024
Sampling Method: Non-Probability Sample
Enrollment: 728 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative 30-day morbidity rate | From enrollment to the postoperative day 30
  • To determine whether preoperative anemia is associated with increased risk of postoperative 30-day morbidity in patients undergoing liver resection.

SECONDARY OUTCOMES:
Allogenic blood transfusion, comprehensive complication index, postoperative outcomes, and mortality rate | From enrollment to the postoperative day 30
  * To determine the incidence of preoperative anemia in liver resection patients.
  * To determine the incidence of postoperative 30-day morbidities rate
  * To evaluated the postoperative 30-day morbidities rate, classified using:
    * Clavien Dindo classification
    * Comprehensive complication index (CCI)
  * To determine postoperative major complication, defined as Clavien-Dindo classification grade III or higher or CCI > 40
  * To assess the length of hospital stay
  * To assess the length of ICU stay and ventilator day
  * To evaluate postoperative 30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Warangkana Lapisatepun, MD. PhD., Principal Investigator — Chiang Mai University

IPD SHARING:
Plan to Share IPD: No